CLINICAL TRIAL: NCT04040725
Title: Phase II Clinical Trial of Rogaratinib for High Risk Non-Muscle Invasive Bladder Cancer (NMIBC) Unresponsive to Bacillus Calmette-Guerin (BCG) With FGFR1 or FGFR3 Gene Overexpression: The Bladder Cancer Signal Seeking Trial (BLASST)-3
Brief Title: Rogaratinib for BCG Refractory High Risk Non-Muscle Invasive Bladder Cancer With FGFR1/2 Overexpression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn per Bayer
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Bradley A. McGregor, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-205
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Rogaratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rogaratinib (Experimental): * Rogaratinib is administered orally twice daily
  * Rogaratinib is held for 72 hours before cystoscopy/TURBT and if no complications are seen, treatment is resumed 24 hours after the TURBT
  Interventions: Drug: Rogaratinib

INTERVENTIONS:
Drug: Rogaratinib — Rogaratinib is an oral drug that inhibits FGFR. Mutations in FGFR help bladder cancer grow.

SUMMARY:
This research study is studying the safety, tolerability, and tumor activity of the study drug known as rogaratinib as a possible treatment for bladder cancer.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied. The U.S. Food and Drug Administration (FDA) has not approved rogaratinib as a treatment for any disease.

In this research study, the investigators are studying rogaratinib in bladder cancer that has not responded to BCG and overexpresses a protein called FGFR1 or 3.

* Mutations in FGFR help bladder cancer grow. In metastatic cancers that express FGFR 1 or 3, rogaratinib and other inhibitors of FGFR have shown to be an effective treatment
* Rogaratinib is an oral drug that inhibits FGFR
* To date, no therapy has been shown to be effective in controlling bladder cancer after BCG does not work.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age (at least age of legal maturity)
* Have a histologically-confirmed diagnosis of high risk non-muscle-invasive (T1, High Grade Ta and/or CIS) transitional cell carcinoma of the bladder. Subjects with tumors of mixed transitional/non-transitional cell histology are not allowed.
* In subjects with Ta and T1, have undergone complete TURBT as characterized by:

  * Attainment of a visually complete resection
  * Residual CIS not amenable to complete transurethral resection is acceptable
  * The most recent cystoscopy / TURBT must have been performed within 8 weeks prior to the first dose of trial treatment
* Have been treated with adequate BCG therapy and have developed NMIBC that is unresponsive to BCG therapy. Adequate BCG therapy must include: An induction course with at least 5 instillations of BCG (adequate induction); and at least 7 instillations of BCG within 9 months of the first instillation of adequate induction therapy. BCG unresponsive high risk NMIBC is defined as: Stage progression at 3 months (±4 weeks) despite adequate induction therapy (e.g., Ta to T1, or CIS to T1; note: adequate induction therapy only, defined above, is required in this case); or Persistent high risk NMIBC at 6 months (±4 weeks) after adequate BCG therapy or Recurrent high risk NMIBC within 9 months of the last BCG instillation despite adequate BCG therapy.
* Have elected not to undergo, or are considered ineligible for radical cystectomy, as determined by the treating surgeon. Reasons for ineligibility or refusal of radical cystectomy should be discussed with the subject as part of the informed consent process and should be captured on the appropriate case report form. Ineligibility factors for radical cystectomy may include, but are not limited to:

  * Cardiovascular disease (e.g. recent acute coronary syndrome, arrhythmia, heart failure)
  * Chronic obstructive pulmonary disease that would preclude a safe surgical procedure, as determined by the treating surgeon
  * Poor performance status (e.g. ECOG >2)
  * Prior major abdominal and pelvic surgery, that would preclude a safe surgical procedure, as determined by the treating surgeon
* High FGFR 1/3 mRNA expression levels (RNAscope score of 3+ or 4+; measurement is part of the protocol) in archival or fresh tumor biopsy specimen
* Existence of archival or fresh tumor biopsy specimen for FGFR1/3 mRNA expression testing. Patients who don't have archival tissue specimens meeting eligibility requirements may undergo a biopsy. Acceptable samples include core needle biopsies for deep tumor tissue (minimum three cores) or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions.
* Ability to understand and signing of the written patient information/informed consent form (PI/ICF) for FGFR testing
* Ability to understand and signing of the written PI/ICF for study treatment eligibility. Signed informed consent form must be available before any study-specific procedure for the respective study parts may begin.(PI/ICF for study treatment eligibility must be offered only after positive results in FGFR testing study received by site.)
* Eastern Cooperative Oncology Group performance status 0 or 1
* Adequate bone marrow, liver and renal function as assessed by laboratory requirements conducted within 14 days before registration:

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3 (without granulocyte colony-stimulating factor support within 2 weeks before the first study drug administration)
  * Hemoglobin ≥ 10 g/dL (without transfusion or erythropoietin within 4 weeks before the first study drug administration)
  * Platelet count ≥ 100,000/mm3 (without transfusion within 2 weeks before the first study drug administration)
  * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN). Total bilirubin ≤ 3 x ULN for patients with known Gilbert syndrome.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
  * Alkaline phosphatase ≤ 2.5 times ULN
  * Lipase and amylase ≤ 2 x ULN
  * Serum albumin ≥ 2.5 g/dl
  * Glomerular filtration rate (GFR) ≥ 40 mL/min/1.73 m2 according to the modification of diet in renal disease (MDRD) abbreviated formula.

Note: at the investigator's discretion, an estimated creatinine clearance result <60 mL/min/1.73m² may be verified by measurement of creatinine clearance based on 24-hour urine collection or using EDTA, inulin, GFR scan. INR ≤ 1.5 x ULN and PTT or activated PTT (aPTT) ≤ 1.5 x ULN. Patients being treated with anticoagulant, e.g. warfarin or heparin, will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists and they are on a stable dose as defined by the local standard of care.

* Negative serum pregnancy test in women of childbearing potential (performed within 7 days before the first treatment). Negative results must be available before the first study drug administration. Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the informed consent form and until at least 5 months after the last study drug administration. The definition of adequate contraception will be based on the judgment of the investigator and on local requirements. Acceptable methods of contraception include, but are not limited to, (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception.
* Recovery to National Cancer Institute's Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v.5.0) Grade 0 or 1 level or recovery to baseline preceding the prior treatment from any previous drug / procedure-related toxicity (patients with persistent alopecia of any grade, and/or anemia [hemoglobin ≥ 10 g/dL] can be included)

Exclusion Criteria:

* Has muscle invasive (i.e. T2, T3, T4) locally advanced non-resectable or metastatic urothelial carcinoma.
* Has concurrent extra-vesical (i.e. urethra, ureter or renal pelvis) non-muscle invasive transitional cell carcinoma of the urothelium.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has undergone any intervening intravesical chemotherapy or immunotherapy from the time of most recent cystoscopy/TURBT to starting trial treatment. (Note: intravesical treatment given as part of the most recent cystoscopy / TURBT is allowed.)
* Previous treatment with anti-FGFR directed therapies (e.g. receptor tyrosine kinase inhibitors including rogaratinib or FGFR-specific antibodies).
* Previous or concurrent cancer except: cervical carcinoma in situ, treated basal-cell carcinoma or squamous cell skin cancer, localized prostate cancer treated with curative intent and known absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (T1/T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL undergoing active surveillance and treatment-naïve), or any other cancer curatively treated > 3 years before the first study drug administration.
* History or current condition of an uncontrolled cardiovascular disease including any of the following conditions:

  * Congestive heart failure (CHF) NYHA Class 2 or greater, unstable angina (symptoms of angina at rest)
  * New-onset angina (within last 3 months before the first study drug administration)
  * Myocardial infarction (MI) within past 6 months before the first study drug administration
  * Unstable cardiac arrhythmias requiring anti-arrhythmic therapy. Patients with arrhythmia not requiring therapy or under control with anti-arrhythmic therapy such as beta-blockers or digoxin are eligible.
* Patients with known coronary artery disease, or congestive heart failure not meeting the above criteria, must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Known human immunodeficiency virus (HIV) infection.
* Active hepatitis B virus (HBV; chronic or acute; defined as having a known positive hepatitis B surface antigen [HBsAg] test at the time of screening) or hepatitis C infection requiring treatment. Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible if HBV DNA is negative. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Active tuberculosis.
* Treatment with therapeutic oral or I.V. antibiotics within 2 weeks before the first study drug administration. Patients receiving prophylactic antibiotics (e.g. for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
* Any hemorrhage / bleeding event CTCAE v.5.0 ≥ Grade 3 within 4 weeks before the first study drug administration.
* Serious, non-healing wound, ulcer, or bone fracture.
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
* Any malabsorption condition.
* Current diagnosis of any retinal disorders including retinal detachment, retinal pigment epithelial detachment (RPED), serous retinopathy or retinal vein occlusion. An ophthalmological exam with optical coherence tomography is required within 30 days of the date of registration.
* Peripheral sensory neuropathy of CTCAE v.5.0 Grade 2 or higher.
* Current evidence of endocrine alteration of calcium phosphate homeostasis (e.g. parathyroid disorder, history of parathyroidectomy, tumor lysis, tumoral calcinosis, paraneoplastic hypercalcemia).
* Concomitant therapies that are known to increase serum phosphate levels (i.e. antacids, laxatives oral/rectal, oral phosphate binders, potassium phosphate) and that cannot be discontinued or switched to a different medication before the first study drug administration.
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.
* Clinically active infections (CTCAE v. 5.0 ≥ Grade 1) within 2 weeks before the first study drug administration.
* Seizure disorder requiring medication.
* History of organ allograft.
* Evidence or history of bleeding diathesis or coagulopathy.
* Women who are actively breastfeeding.
* Use of strong inhibitors of CYP3A4 and strong inducers of CYP3A4 are not permitted for 2 weeks before the first study drug administration or during the study.
* Autologous bone marrow transplant or stem cell rescue within 4 months before the first study drug administration.
* Major surgery, open biopsy, or significant traumatic injury within 4 weeks before the first study drug administration (central line surgery is not considered major surgery).
* Renal failure requiring peritoneal dialysis or hemodialysis.
* Systolic/diastolic blood pressure ≤ 100/60 mmHg and concurrent heart rate ≥ 100/min.
* Inability to swallow oral tablets.
* Close affiliation with the investigational site; e.g. a close relative of the investigator or a dependent person (e.g. employee of or student at the investigational site).
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Arterial or venous thrombotic events or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the first study drug administration.
* Those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Concomitant therapy with the following medication is prohibited

  * Concomitant use of strong inhibitors of CYP3A4 and strong inducers of CYP3A4 are not permitted for 2 weeks prior to start of study treatment or during the study.
  * Concomitant use of moderate and weak CYP3A4 inducers should be avoided as clinically significant decrease in plasma concentrations of rogaratinib cannot be ruled out.
  * Concomitant use of herbal preparations containing CYP3A4 inducers (e.g. St John's Wort) are not permitted during the study.
  * Grapefruit and grapefruit juice (CYP3A4 inhibitor) consumption is not permitted during the study.
  * Therapies that are known to increase serum calcium or phosphate levels (i.e. antacids, phosphate-containing laxatives oral/rectal, potassium phosphate)
  * Patients may not receive other investigational treatment or other approved anti-tumor therapy while on this protocol (excluding anti-VEGF therapy for ophthalmologic disease).
* Concomitant therapies that should be avoided:

  * Narrow therapeutic index drugs that are CYP3A4, P-gp, and BCRP substrates (e.g. alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, and tacrolimus) should be avoided, because drug interactions caused by irreversible inhibition of CYP3A4, P-gp, and BCRP by rogaratinib cannot be ruled out.
  * Fluconazole is considered a moderate to strong inhibitor of CYP2C9 and should be avoided, if possible.
  * No results are available from human interaction studies between rogaratinib and other chemotherapies. No data are available to evaluate the interaction between rogaratinib and radiation. Therefore, when administering these agents after study drug has been withdrawn, it should be taken into consideration that rogaratinib plasma concentrations may be detectable for a few days (depending on half-life) and the physiologic consequences that could interact with chemotherapy and radiotherapy may last even longer following discontinuation of rogaratinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Complete Response | 6 months
  Absence of any cancer in the bladder (No carcinoma in situ or new lesions) on examination with TURBT

SECONDARY OUTCOMES:
Duration of Response | 2 years
  Duration of time from study entry until appearance of any cancer in the bladder (No carcinoma in situ or new lesions) on examination with TURBT
Rate Toxicity Occurs | 2 years
  Percentage of patients with a side effect from rogaritinib while on study

CONTACTS AND LOCATIONS:
Overall Officials: Bradley A. McGregor, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu